CLINICAL TRIAL: NCT06324097
Title: Diagnostic Value of Two Different Mode Endocytoscopy for Colorectal Lesions
Brief Title: Diagnostic Value of Endocytoscopy for Colorectal Lesions
Status: Completed | Type: Observational
Sponsor: Hong Xu (Other)
Responsible Party: Sponsor-Investigator, Hong Xu, Director, Head of Gastroenterology and Endoscopy Center, Principal Investigator, Clinical Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: 2024-623
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Post-operative colorectal lesion specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal lesion
  Interventions: Diagnostic Test: endocytoscopy

INTERVENTIONS:
Diagnostic Test: endocytoscopy — The colorectal lesions had been observed with EC-NBI and EC-stained by endoscopists before treatment that were ultimately performed histopathologic examination. The endocytoscopies (CF-H290ECI, Olympus, Tokyo, Japan) have a maximum magnification of ×520, focusing depth, 35 μm; field of view, 570 × 500μm. During EC-NBI , the endoscopist pushed the button of the endoscope to switch from white-light imaging to NBI and observed the lesion with full magnification. Finally, the endoscopist performed EC-stained mode diagnosis after staining the lesion surface with 1.0% methylene blue.

SUMMARY:
Colorectal cancer (CRC) is the third most common malignancy and the second leading cause of cancer-related death worldwide. Colonoscopy is considered the preferred method of screening for colorectal cancer, and resection of colorectal lesions can significantly reduce the incidence and mortality of colorectal cancer. In order to improve the qualitative and quantitative diagnosis of colorectal lesions, many endoscopic techniques, such as image-enhanced endoscopy (IEE), including narrowband imaging (NBI), magnifying endoscopy, pigment endoscopy, confocal laser endoscopy, and endocytoscopy (EC) are applied clinically. The application of EC is intended to achieve the purpose of real-time histopathological endoscopic diagnosis without biopsy. Several studies have shown that EC is effective in identifying the nature of colorectal lesions and judging the depth of invasion in CRC. Based on the endoscopic diagnosis, the endoscopist can determine the treatment plan for the colorectal lesions. The latest EC is an integrated endoscope with a contact light microscopy system with a maximum magnification of 520 x. EC may demonstrate the atypical of gland structure and cells after staining (EC staining mode, along with the use of the EC-NBI mode. The endoscopic diagnosis of the EC staining mode is based on the EC classification (EC-C), used to predict the histopathological diagnosis of colorectal lesions. A prospective randomized trial showed that the diagnostic accuracy was 94.1% by EC-C. However, the diagnostic value of EC-C depends on the operator and may be influenced by the quality of the staining. Meanwhile, the high-quality staining process is time-consuming and tedious. Therefore, EC-NBI seems to be the first choice for EC diagnosis with the advantages of convenient operation and efficient diagnosis. EC-NBI can display the super-amplified surface microvessels of the lesion and provide pathological prediction according to the vessel classification (EC-V). EC-V achieved 99% diagnostic accuracy for hyperplastic polyps and 88.6% for invasive carcinoma. In EC examination, the investigators usually use EC-NBI and EC staining successively to diagnose colorectal lesions, which is believed to improve the diagnostic performance. However, the diagnostic value of increasing EC-staining after EC-NBI examination for predicting the pathological nature of colorectal lesions is still unclear. Therefore, this retrospective study aimed to evaluate the diagnostic value of two different modalities of cell endoscopy for colorectal lesions and to clarify whether additional EC staining after EC-NBI could improve the diagnostic performance of predicting the pathological diagnosis of colorectal lesions.

In the study, the investigators collect clinical information of colorectal lesions which were diagnosed by endoscopic diagnosis (including EC-NBI and EC-staining) and pathological diagnosis. Then, the investigators calculate the accuracy, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and high confidence diagnosis rate of EC-C and EC-V classification, respectively. Inter-and intra-observer agreement in the diagnosis of EC-C and EC-V will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* colorectal lesions

Exclusion Criteria:

* non-epithelial tumors
* sessile serrated lesions
* inflammatory polyps
* juvenile polyps
* hamartomatous polyps
* a history of inflammatory bowel disease
* chemotherapy or radiation therapy for colorectal cancer
* lesions without clear EC images.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators analyzed only endoscopically or surgically resected colorectal lesions (hyperplastic polyps, adenomas and invasive cancers) that had been observed with EC-NBI and EC-stained by endoscopists before treatment that were ultimately performed histopathologic examination.
Sampling Method: Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
sensitivity | April 2024
specificity | April 2024
accuracy | April 2024
positive predictive value | April 2024
negative predictive value | April 2024

SECONDARY OUTCOMES:
inter-observer agreement | April 2024
intra-observer agreement | April 2024

CONTACTS AND LOCATIONS:
Locations (1):
- the Department of Gastroenterology and Endoscopy Center, First Hospital of Jilin University, Changchun, Jilin, China